CLINICAL TRIAL: NCT02711176
Title: Comparison of Daily Single Dose Triple and Conventional Triple Therapies for Helicobacter Pylori Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zahra Vahdat Shariatpanahi (Other)
Responsible Party: Sponsor-Investigator, Zahra Vahdat Shariatpanahi, Assistant Professor, Ilam University of Medical Sciences
Organization: Ilam University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22/52/1662
Record Dates: First submitted 2016-02-09; First posted 2016-03-17 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Helicobacter Infection
MeSH Terms: conditions — Helicobacter Infections | interventions — Esomeprazole; Tinidazole; Lansoprazole; Clarithromycin; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (2):
- Tavanex & Nexium & Tinafas (Experimental): Patients will receive Nexium (Esomeprazole) 40 mg daily and Tinafas (Tinidazole) 1 g daily and Tavanex (Levofloxacin) 500 mg daily for 14 days"
  Interventions: Drug: Nexium; Drug: Tinafas; Drug: Tavanex
- Lanzol & Klacid &Iramox (Active Comparator): Patients will receive Lanzol (lansoprazole) 30 mg twice daily and Klacid (clarithromycin) 500 mg twice daily and Iramox (amoxicillin) 1 g twice daily for 14 days
  Interventions: Drug: Lanzol; Drug: Klacid; Drug: Iramox

INTERVENTIONS:
Drug: Nexium — Patients in experimental group will receive the 14 day single dose of Nexium 40 mg daily
  Other Names: Esomeprazole
  Arms: Tavanex & Nexium & Tinafas
Drug: Tinafas — Patients in experimental group will receive the 14 day single dose regimen of Tinafas 1 g daily
  Other Names: Tinidazole
  Arms: Tavanex & Nexium & Tinafas
Drug: Tavanex — Patients in experimental group will receive the 14 day single dose of Tavanex 500 mg daily
  Other Names: Levofluxacine
  Arms: Tavanex & Nexium & Tinafas
Drug: Lanzol — Patients in active comparator group will receive the 14 day lansoprazole (Lanzol) 30 mg twice daily
  Other Names: lansoprazole
  Arms: Lanzol & Klacid &Iramox
Drug: Klacid — Patients in active comparator group will receive the 14 day clarithromycin (Klacid) 500 mg twice daily twice daily
  Other Names: clarithromycin
  Arms: Lanzol & Klacid &Iramox
Drug: Iramox — Patients in active comparator group will receive the 14 day amoxicillin (Iramox) 1 g twice daily
  Other Names: amoxicillin
  Arms: Lanzol & Klacid &Iramox

SUMMARY:
This study is conducted to investigate whether the efficacy of single-dose triple therapy (Esomeprazole 40 mg, Tinidazole 1 g, and Levofluxacine 500 mg) for 14 days is superior to double-dose lansoprazole 30 mg, amoxicillin 1 g and clarithromycin 500 mg for 14 days in the treatment of H pylori infection.

DETAILED DESCRIPTION:
Multiple regimens have been evaluated for H. pylori therapy in randomized controlled trials The treatment regimen that is selected must be effective, but considerations such as cost, side effects, and ease of administration should also be taken into account. Despite the number of studies, the optimal therapeutic regimen has not yet been defined.

The regimen most commonly recommended for first line treatment of H. pylori is triple therapy with a PPI, amoxicillin and clarithromycin for 14 days. However, the multi-drug application is associated with remarkable side effects and it is not uncommon not to be able to complete a treatment course. Thus, treatment failure is associated with H. pylori strains that are resistant to the commonly used antibiotics. This study is conducted to investigate whether the efficacy of single-dose triple therapy (Esomeprazole 40 mg, Tinidazole 1 g, and Levofluxacine 500 mg) for 14 days is superior to double-dose lansoprazole 30 mg, amoxicillin 1 g and clarithromycin 500 mg for 14 days in the treatment of H pylori infection.

ELIGIBILITY:
Inclusion Criteria:

* The patients who proved H. pylori infection following three methods

  * Positive rapid urease test
  * Histologic evidence of H. pylori by modified Giemsa staining
  * Positive stool Antigen Test

Exclusion Criteria:

* Patients who received eradication therapy for H. pylori infection, previously
* H. pylori eradication failure because of poor compliance
* The administration of antibiotics or the consumption of bismuth salts within 4 weeks or the administration of a proton pump inhibitor (PPI) within 2 weeks
* Advanced gastric cancer or other malignancy
* Abnormal liver function or liver cirrhosis
* Abnormal renal function or chronic kidney disease
* Other severe concurrent diseases
* Previous allergic reactions to the study drugs
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2016-09; Primary Completion 2017-03-27 (Actual); Study Completion 2017-03-27 (Actual)

PRIMARY OUTCOMES:
The rate of H.pylori eradication | 42 days after study completion
  Breath Urea Test

SECONDARY OUTCOMES:
Drug Compliance | within the first week after study completion
  Interview

CONTACTS AND LOCATIONS:
Overall Officials: Shaahin Shahbazi, MD, Principal Investigator — Assistant Professor, Ilam University of Medical Sciences,Head of Faculty of Medicine
Locations (1):
- Ilam University of Medical Scienvc, Īlām, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shahbazi S, Vahdat Shariatpanahi Z. Comparison between daily single-dose triple therapy and conventional triple therapy on patient compliance and Helicobacter pylori eradication: A randomized controlled trial. Indian J Gastroenterol. 2018 Nov;37(6):550-554. doi: 10.1007/s12664-018-0916-z. Epub 2019 Jan 12. PMID 30635887